CLINICAL TRIAL: NCT04878172
Title: Histological Study to Assess Safety and Efficacy of the TempSure Firm for Non-Invasive Lipolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7027-MCPL-2021
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Results first posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Non-invasive Lipolysis

STUDY DESIGN:
Intervention Model Description: There are 4 different arms, each with different time frames based on thei subjects' availability. Each group uses the same device and treatment parameters, with the only difference being when follow up measures are taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- TempSure Firm Day 0 Biopsy Group (Experimental): Subjects will undergo abdominal surgery after an abdominal treatment with TempSure Firm at day 0 (within 24 hours after treatment).
  Interventions: Device: TempSure Firm
- TempSure Firm Day 10 Biopsy Group (Experimental): Subjects will undergo abdominal surgery after an abdominal treatment with TempSure Firm at day 10 (+/- 3 days) after treatment.
  Interventions: Device: TempSure Firm
- TempSure Firm Day 20 Biopsy Group (Experimental): Subjects will undergo abdominal surgery after an abdominal treatment with TempSure Firm at day 20 (+/- 3 days) after treatment.
  Interventions: Device: TempSure Firm
- TempSure Firm Day 30 Biopsy Group (Experimental): Subjects will undergo abdominal surgery after an abdominal treatment with TempSure Firm at day 30 (+/- 7 days) after treatment.
  Interventions: Device: TempSure Firm

INTERVENTIONS:
Device: TempSure Firm — The TempSure firm will be used on the abdomen for non-invasive lipolysis.

SUMMARY:
This is a prospective, open-labeled, non-randomized, multi-center clinical study to collect safety and efficacy data on the TempSure Firm. The intended use of the TempSure device is to use the Firm handpieces for non-invasive lipolysis.

DETAILED DESCRIPTION:
Up to 12 subjects will be enrolled at up to 3 study centers. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive 1 treatment on the abdomen with the TempSure firm. Subjects will undergo abdominoplasty surgery at one of 4 predetermined timepoint after an abdomen treatment: day 0 (within 24 hours after treatment), 10 days (+/- 3 days), 20 days (+/- 3 days), or 30 days (+/- 7 days). This will be determined by the availability of the subject and/or an as needed basis and this will be decided by the Investigator and the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 - 55 years old.
* Willing to receive treatments with the TempSure® device and willing to have biopsies taken from a control site and the treatment area (biopsies are collected after the abdominal tissue flap is removed during abdominoplasty surgery)
* Understand and accept obligation not to receive any other procedures on the treatment and control areas throughout the length of the study.
* Understand and accept the obligation and able to be present for all study visits
* Willing to comply with all requirements of the study and able to provide informed consent.

Exclusion Criteria:

Pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning to become pregnant prior to the end of the study.

* Currently enrolled in an investigational drug or device trial, or has received an investigational drug or investigational device treatment(s) in the area to be treated (or designated control area) 6 months prior to entering this study (or at the discretion of the Investigator) .
* Cuts, wounds, or infected skin on the area to be treated or designated control area
* On local, oral, or systemic anesthetic agents.
* Condition(s) or circumstance(s) that, in the investigators opinion, may put the subject at significant risk, may confound study results or may interfere significantly with subject participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (2):
- United States (2):
  - Bass Plastic Surgery PLLC, New York, New York
  - Aesthetic Pavilion Ambulatory Surgery Center, Staten Island, New York

REFERENCES:
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TempSure Firm Day 0 Biopsy Group | TempSure Firm Day 10 Biopsy Group | TempSure Firm Day 20 Biopsy Group | TempSure Firm Day 30 Biopsy Group
Started | 2 | 2 | 2 | 3
Completed | 2 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TempSure Firm Day 0 Biopsy Group | TempSure Firm Day 10 Biopsy Group | TempSure Firm Day 20 Biopsy Group | TempSure Firm Day 30 Biopsy Group | Total
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 3 | 9
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 3 | 8
  Male | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 0 | 0 | 1 | 1
  Caucasian | 2 | 2 | 2 | 2 | 8
FitzPatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is. The scale comes from the source listed in the references.
  Participants
    Fitzpatrick Skin Type I | 0 | 0 | 0 | 0 | 0
    Fitzpatrick Skin Type II | 0 | 1 | 0 | 1 | 2
    Fitzpatrick Skin Type III | 1 | 1 | 2 | 1 | 5
    Fitzpatrick Skin Type IV | 1 | 0 | 0 | 0 | 1
    Fitzpatrick Skin Type V | 0 | 0 | 0 | 1 | 1
    Fitzpatrick Skin Type VI | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Histology of Biopsy
Description: Subjects will undergo abdominal surgery after an abdominal treatment with TempSure Firm within 24 hours post treatment. The samples were looked at from a qualitative standpoint to determine of whether the samples had signs of adipocyte injury and/or inflammatory tissue response, and if there was dermal/epidermal tissue injury (which was assessed by a qualified histologist).
Time Frame: within 24 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | TempSure Firm Day 0 Biopsy Group
Number analyzed (Participants) | 2
Participants
  # of participants whose sample had signs of adipocyte injury and/or inflammatory tissue response. | 2
  # of participants whose sample had no epidermal or dermal tissue injury | 2

2. Primary Outcome: Histology of Biopsy
Description: Subjects will undergo abdominal surgery after an abdominal treatment with TempSure Firm at day 10 (+/- 3 days) after treatment. The samples were looked at from a qualitative standpoint to determine of whether the samples had signs of adipocyte injury and/or inflammatory tissue response, and if there was dermal/epidermal tissue injury (which was assessed by a qualified histologist).
Time Frame: within 10 days (+/- 3 days) post treatment
Measure: Number; unit: participants
Arm/Group | TempSure Firm Day 10 Biopsy Group
Number analyzed (Participants) | 2
participants
  # of participants whose sample had signs of adipocyte injury and/or inflammatory tissue response. | 2
  # of participants whose sample had no epidermal or dermal tissue injury | 2

3. Primary Outcome: Histology of Biopsy
Description: Subjects will undergo abdominal surgery after an abdominal treatment with TempSure Firm at day 20 (+/- 3 days) after treatment. The samples were looked at from a qualitative standpoint to determine of whether the samples had signs of adipocyte injury and/or inflammatory tissue response, and if there was dermal/epidermal tissue injury (which was assessed by a qualified histologist).
Time Frame: within 20 days (+/- 3 days) post treatment
Measure: Number; unit: participants
Arm/Group | TempSure Firm Day 20 Biopsy Group
Number analyzed (Participants) | 2
participants
  # of participants whose sample had signs of adipocyte injury and/or inflammatory tissue response. | 2
  # of participants whose sample had no epidermal or dermal tissue injury | 2

4. Primary Outcome: Histology of Biopsy
Description: Subjects will undergo abdominal surgery after an abdominal treatment with TempSure Firm at day 30 (+/- 3 days) after treatment. The samples were looked at from a qualitative standpoint to determine of whether the samples had signs of adipocyte injury and/or inflammatory tissue response, and if there was dermal/epidermal tissue injury (which was assessed by a qualified histologist).
Time Frame: within 30 days (+/- 7 days) post treatment
Measure: Number; unit: participants
Arm/Group | TempSure Firm Day 30 Biopsy Group
Number analyzed (Participants) | 3
participants
  # of participants whose sample had signs of adipocyte injury and/or inflammatory tissue response. | 3
  # of participants whose sample had no epidermal or dermal tissue injury | 3

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) occurring were captured and followed up throughout the study duration, approximately 2 months.
Arm/Group | TempSure Firm Day 0 Biopsy Group | TempSure Firm Day 10 Biopsy Group | TempSure Firm Day 20 Biopsy Group | TempSure Firm Day 30 Biopsy Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT04878172/Prot_SAP_000.pdf